CLINICAL TRIAL: NCT00442728
Title: on Muscle Wasting in Artificially Ventilated and Sedated Patients at the Intensive Care Unit: a Pilot Study
Brief Title: The Effect of Neuromuscular Electrical Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Provinciale Hogeschool Limburg (Other)
Collaborators: KU Leuven (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REVAL300107
Record Dates: First submitted 2007-02-11; First posted 2007-03-02 (Estimated); Last update posted 2007-03-02 (Estimated); Status verified 2007-03

CONDITIONS: Postoperative Coronary Artery Bypass Grafting (CABG); Chronic Obstructive Pulmonary Disease (COPD); Ventilatory Failure
Keywords: Functional electrical stimulation; muscular atrophy; intensive care
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoventilation; Muscular Atrophy | interventions — Electric Stimulation

INTERVENTIONS:
Device: ELECTRICAL STIMULATION

SUMMARY:
The effect of neuromuscular electrical stimulation on muscle atrophy in sedated patients on intensive care was studied. The aim of this study was to explore if electrical stimulation could prevent muscle atrophy.

DETAILED DESCRIPTION:
Patients were included in the study one day after administration when prolonged sedation and ventilation were expected. They were divided into intervention (n=7) and control (n=14) groups. For the intervention group, an intermittent neuromuscular electrical stimulation was applied daily for 30 minutes on the right thigh whereas the left thigh was used as a control. Heart rate, respiration rate, systolic and diastolic blood pressure and oxygen saturation were monitored before, during and after the electrostimulation. Perimeter of the right and left thighs was measured in both groups every 3 days at 5 cm above the upper edge of the kneecap.

ELIGIBILITY:
Inclusion Criteria:

* . Prior to inclusion in the study, an informed consent was given by the family of the patients which was approved by the local Ethics Committee of the Virga Jesse Hospital and was performed in accordance with the standards of the 1964 Declaration of Helsinki.

Exclusion Criteria:

* Patients were excluded from the study if they were still able to move their limb actively in spite of the sedation. Patients were also excluded if they had signs of recent ischemia or infarction for less then seven days. Patients with severe orthopaedic or vascular damage, i.e., fractures or oedema in the lower limbs were also excluded. Patients with an augmented risk for neuro electrical stimulation such as open wounds, hemodialysis or an arterial catheter at the stimulation area were also excluded.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21
Dates: Start 2003-01; Study Completion 2003-06

PRIMARY OUTCOMES:
Perimeter of the right and left thighs was measured in both groups every 3 days at 5 cm above the upp

CONTACTS AND LOCATIONS:
Overall Officials: RAf LJ Meesen, Phd, Principal Investigator — PHL
Locations (1):
- REVAL, Hasselt, LIMBURG, Belgium